CLINICAL TRIAL: NCT02167503
Title: A Retrospective-prospective Observational Study to Evaluate the Effect of Anti-viral Treatment on the Long-term Outcome in Patients With Chronic Hepatitis B (SEARCH-B Study)
Brief Title: Observational Study on Patients With Chronic Hepatitis B
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: National Health and Family Planning Commission, P.R.China (Other Government)
Responsible Party: Sponsor
Other Study IDs: MOH-08
Record Dates: First submitted 2014-06-17; First posted 2014-06-19 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study was conducted to evaluate the effect of anti-viral treatment on long-term outcome on patients with chronic hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged over 30 (inclusive) years of old
* Patients has a history of diagnosis of chronic hepatitis B (ie. HBsAg positive for more than 6 months)
* For patients with HBsAg positive, patients should be undergoing anti-viral treatment
* For patients with HBsAg negative, a documented evidence of previous anti-viral treatment should be provided.
* Life expectancy is more than 1 year
* Good treatment compliance.

Exclusion Criteria:

* Patients has a history of diagnosis of hepatocellular carcinoma
* Patients with Child Pugh C
* Coinfected with HCV, HDV and HIV
* Suffering from other serious disease
* Taking part in other clinical trial

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis B from hospital
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2014-05; Primary Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Cumulative rates of hepatocellular carcinoma | Year 5

CONTACTS AND LOCATIONS:
Overall Officials: Jinlin Hou, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (14):
- China (14):
  - Beijing Ditan Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital Attached to the Capital Medical University, Beijing, Beijing Municipality
  - BeiJing YouAn Hospital ,Capital Medical University, Beijing, Beijing Municipality
  - Department of infectious disease, First Hospital of Peking University, Beijing, Beijing Municipality
  - People's Hospital of Beijing University, Beijing, Beijing Municipality
  - Department of infectious disease, Nanfang Hospital, Guangzhou, Guangdong
  - The Third Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital Central-South Univrsity, Changsha, Hunan
  - First Hospital .Jilin Unniversity, Changchun, Jilin
  - ShengJing Hospital of China Medical University, Shenyang, Liaoning
  - Huashan Hospital，Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of College of Medicine ，Zhejiang University, Hangzhou, Zhejiang